CLINICAL TRIAL: NCT04091022
Title: A Randomized, Placebo-controlled, Double-blind, Phase II Chemoprevention Clinical Trial of Topical Diclofenac and DFMO in Subjects With a History of Skin Cancer
Brief Title: Topical Diclofenac and Topical DFMO Chemoprevention Trial in Subjects With a History of Skin Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Craig Elmets, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 300004144; R01CA193885 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Non-melanoma Skin Cancer
Keywords: topical chemoprevention
MeSH Terms: interventions — Diclofenac; Eflornithine

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial will be double-blinded. The clinical team and patient will remain blinded to the randomization.
  All study drug will be blinded except to the pharmacists. Records will be kept to document receipt, distribution and disposition of the drugs. Unblinding will only be done at the end of the study or as medically indicated with consent of the study PI and the biostatistician, after consulting the NIH Project Officer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diclofenac + DFMO (Active Comparator): Participants in this arm will apply topical diclofenac to bilateral forearms once per day and topical DFMO to bilateral forearms once per day.
  Interventions: Drug: Solaraze and Vaniqa
- Placebo + Placebo (Placebo Comparator): Participants in this arm will apply placebo for topical diclofenac to bilateral forearms once per day and placebo for topical DFMO to bilateral forearms once per day.
  Interventions: Drug: Solaraze and Vaniqa

INTERVENTIONS:
Drug: Solaraze and Vaniqa — Solaraze-topical diclofenac 3% and Vaniqa-topical eflornithine hydrochloride Cream, 13.9% applied to bilateral arms for a period of 9 months
  Other Names: Solaraze-topical diclofenac 3% and Vaniqa-topical eflornithine hydrochloride Cream, 13.9%

SUMMARY:
This is a single institution, randomized, placebo-controlled, double-blind phase IIB trial of 1) topical diclofenac and topical DFMO, or 2) placebo in participants with a history of non melanoma skin cancer/ keratinocytic cancers.

DETAILED DESCRIPTION:
There will be two groups to the study. Individuals, aged 18 years or older, who have extensive actinic damage, at least 8 AKs and a history of at least one non-melanoma skin cancer, but are in otherwise general good health, will be given topical diclofenac and topical DFMO. They will be compared to individuals, aged 18 years or older, who have extensive actinic damage, but are in otherwise general good health, will be given placebo. All participants must be at increased risk of non-melanoma skin cancer as evidenced by a history of prior squamous or basal cell skin cancer, ongoing or history of actinic keratoses, and the presence, at baseline, of at least eight actinic keratoses on the face, neck, scalp and arms. Subjects will be randomized to:

1. topical diclofenac once daily and topical DFMO once daily
2. placebo for the topical diclofenac once daily and placebo for the topical DFMO once daily

ELIGIBILITY:
Inclusion Criteria

* Previous treatment for basal or squamous cell skin cancer stage 0-2 and current evidence of at least actinic keratosis on the upper extremities (upper arms, forearms and hands), neck, face or scalp.
* >18 years of age
* Ability to understand and willingness to sign a written informed consent document
* ECOG performance status 0-1
* Willing and able to participate for the full duration of the study
* Willing to abstain from:

  * The application of topical medications including prescription and over the counter preparations (e.g., Topical preparations containing corticosteroids or vitamin A derivatives) to intended treatment areas for the duration of the study. Use of moisturizers/emollients and sunscreens on these areas is allowed.
  * Chronic (defined as > 3 times/week for more than 2 consecutive weeks/year) NSAID and COX-2 inhibitor use (other than cardioprotective doses of aspirin < 100 mg po QD) for the duration of the study
* Normal organ and marrow function defined as laboratory values falling within the specified ranges for the following tests (performed within 365 days of registration)

Hematologic

* WBC >3,000/ul
* Hemoglobin > lower limit of normal
* Platelet count > 100,000/ul

Hepatic

* Total bilirubin < 1.5 X ULN
* AST (SGOT) < 1.5 X ULN
* ALT (SPGT) < 1.5 X ULN Renal
* Serum creatinine < 1.5 X ULN BUN < 1.5 X ULN

  • Females of childbearing potential must:
* Have been using adequate contraception (abstinence, IUD, birth control pills or spermicidal gel with diaphragm or condom) since their last menses
* Have a documented negative urine pregnancy test prior to the first dose of study medication. (Females are not considered to be of childbearing potential if they are at least 1 year post-menopausal or have had a tubal ligation, bilateral oophorectomy or hysterectomy)
* The effects of DFMO and diclofenac on the developing fetus are unknown. Therefore, all females of childbearing potential and all men capable of fathering a child must agree to use adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) for the duration of study participation.

Exclusion Criteria

Any of the following will render a participant ineligible to participate in this study:

* Aspirin >100 mg/day
* Chronic (> 3 times/week for more than a two week period) use of NSAIDs or COX-2 inhibitors
* Current use of topical steroids to intended treatment area (forearms)
* Cryotherapy to intended treatment area (forearms) within the preceding 3 months
* Use of oral or intravenous corticosteroids for more than 2 consecutive weeks

Any of the following in the 4 weeks prior to randomization:

* Major surgery for any indication
* Cytotoxic chemotherapy for any indication (including methotrexate for arthritis)
* Anti-cancer treatment of any type other than for a stage 0-2 non-melanoma skin cancer
* Hormonal therapy for cancer prevention ((treatment with finasteride/dutasteride for BPH does not render a participant ineligible.)
* Radiation therapy

Any of the following in the 6 month prior to randomization to the intended treatment area (forearms):

* Topical medications for the treatment of actinic keratosis or skin cancer (etretinate, 5-FU, imiquimod, ingenol)
* Laser resurfacing, dermabrasion, chemical peel and/or electrodissection ± curettage

  * Any family history of Ornithine diaminotransferase deficiency in a first degree relative
  * Any personal history of:
* Invasive cancer diagnosed or treated within the past 5 years. Participants who have been in remission for >5 years and have not required treatment in the past 5 years may be eligible if a study chair or principal investigator believes there is little to no risk of recurrence.
* Solid organ or bone marrow transplant
* Biopsy proven hepatic cirrhosis
* Keloid formation
* Photosensitivity disorder
* Hypersensitivity or adverse reactions to nonsteroidal anti-inflammatory agents
* Oral DFMO for > 1 month on a prior study
* Any disease that predisposes to NMSC
* An immunodeficiency disorder or the use of an immunosuppressive drug

  • Concurrent use of the following medications or treatments:
* Systemic therapy with psoralens, immunotherapy, or retinoids.
* Cytotoxic chemotherapy for any reason (including methotrexate for arthritis)
* Topical or systemic immunosuppressive therapy

  * Females who are pregnant or lactating. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should notify her study physician immediately.
  * Uncontrolled concurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled symptomatic cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements or other underlying serious medical condition which, in the investigator's opinion might preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Reduction of actinic keratoses | one year (9 months on active, continuous treatment)
  The purpose of the study is to determine whether participants randomized to a combination of two FDA approved topical medications topical diclofenac and topical DFMO have a significant change in incidence of (≥ 50% change, p ≤ 0.05) non-melanoma skin cancers (NMSC) than participants randomized to placebo as assessed by clinical and histopathological evaluation.

SECONDARY OUTCOMES:
Safety assessment | one year (9 months on active, continuous treatment)
  Determination of safety of the combination of topical diclofenac and topical DFMO as compared to placebo using the NCI- Common Terminology Criteria for Adverse Events (CTCAE)
Biomarker assessment | one year (9 months on active, continuous treatment)
  To assess the effect of topical diclofenac and topical DFMO on the following biomarkers in biopsied non-sun exposed skin, skin tissue that has chronic sun damage, and in actinic keratosis skin lesions at 0 and 9 months:
  mRNA expression of Sonic Hedgehog, Hip1, Ptch1, Gli1, Gli2, Gli3, and p53, Prostaglandin E2, Proliferation indices (PCNA, cyclin D1), Apoptosis markers (Tunel staining, Bcl-2, caspase-3), Polyamine concentrations (putrescine, spermidine, spermine)
Biomarker assessment of NMSC | one year (9 months on active, continuous treatment)
  Effect of topical diclofenac and topical DFMO on biomarkers of squamous cell skin cancer and basal cell skin cancer which include mRNA expression of p53,proliferation indices (PCNA, cyclin D1),apoptosis markers (Tunel staining, Bcl-2, caspase-3), andmarkers of epithelial adhesion (E-cadherin)

CONTACTS AND LOCATIONS:
Overall Officials: Craug Elmets, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - UAB Dermatology, Birmingham, Alabama